CLINICAL TRIAL: NCT06671561
Title: Product Surveillance Registry (PSR) Ear, Nose and Throat- PROPEL Drug-Eluting Sinus Stent Family EXTEND Cohort
Brief Title: Product Surveillance Registry; Ear, Nose and Throat - EXTEND Cohort
Status: Withdrawn | Type: Observational
Why Stopped: New study design and data collection needed
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: EXTEND
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Chronic Rhinosinusitis (CRS)
Keywords: PROPEL; Corticosteroid-eluting sinus implants; Product Surveillance Registry ENT; PROPEL Mini; PROPEL Contour

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Observational data collection from patients with chronic rhinosinusitis (CRS) receiving PROPEL sinus implant(s) following functional endoscopic sinus surgery (FESS) — Observational data collection

SUMMARY:
The purpose of this study is to confirm long-term clinical safety and performance, acceptability of identified risks, and detect emerging risks based on factual evidence for the PROPEL family of products when used according to labeling in a real-world setting.

DETAILED DESCRIPTION:
Ongoing clinical investigation for the purpose(s) of:

* Providing continuing evaluation and periodic reporting of safety and effectiveness of Medtronic market-released products for their intended use
* Obtaining real-world performance and safety information from a global network of hospitals, clinics, and clinicians intended to represent the range of clinical environments in which Medtronic products are used
* Supporting post-market surveillance activities and post-approval studies that are initiated by Medtronic, regulated by local governments, or are conducted to fulfill government and/or regulatory authority requests
* Obtaining clinical evidence to guide the development and improvement of medical devices, therapies, device guidelines, and patient services/solutions
* Providing clinical data to support health economics and clinical outcomes research

Enrollment is estimated to take place at up to 10 sites in Europe over 12 months. A single site may enroll no more than 30 patients. Patients may be enrolled up to 60 days prior to the baseline procedure. Subjects will be followed for a total duration of12 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patient or legally authorized representative (LAR) provides authorization and/or consent per institution and geographical requirements.
* Patient has or is intended to receive or be treated with an eligible Medtronic product
* Patient is consented within the enrollment window of the therapy received, as applicable

Exclusion Criteria:

* Patient who is, or is expected to be, inaccessible for follow-up
* Participation is excluded by local law
* Patient is currently enrolled or plans to enroll in concurrent drug/device study that may confound the PSR results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is the European CRS population implanted with Propel implants. Patients included in the analysis population should have a confirmed diagnosis of CRS with or without nasal polyps (NP) and are indicated for FESS (defined as total SNOT-22 score >/= 20 and Lund-Mackay score >/= 1 in each sinus intended to receive an implant. Patients should not have received biologic medication approved for treatment of CRSwNP in </= 12 weeks prior to the baseline FESS procedure, and the FESS procedure should be completed with attempted placement of 1-4 corticosteroid-eluting implants in the ethmoid sinus and/or FSO. Patients should not have had packing materials or splints of any kind placed within the implants unless medically necessary.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-01-30 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
To characterize the SNOT-22 total score change from baseline to Month 6 in patients with CRS undergoing FESS | From baseline (prior to FESS procedure and sinus implant) to 6 months post procedure
  The primary objective is to characterize the Sino-Nasal Outcome Test 22 item (SNOT-22) total score change from baseline to Month 6. The SNOT-22 assesses 22 symptoms associated with Chronic Rhinosinusitis (CRS) with a value from 0 (no problem) to 5 (problem as bad as it can be). The total score is assessed by summing the score for each of the 22 items. Baseline SNOT-22 total scores are expected to be higher prior to Functional Endoscopic Sinus Surgery (FESS) and implant of the sinus implant(s) . A decrease in SNOT-22 score at 6 months would indicate improvement in the patient's CRS symptoms.

IPD SHARING:
Plan to Share IPD: No